CLINICAL TRIAL: NCT02402101
Title: Effect of the Transcranial Direct Current Stimulation on the Dopaminergic
Brief Title: Effect of the Transcranial Direct Current Stimulation on the Dopaminergic Transmission in Healthy Subjects
Acronym: DOPA-STIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2014-A01405-42
Record Dates: First submitted 2015-03-18; First posted 2015-03-30 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Transcranial Direct Current Stimulation; Dopamine
Keywords: tDCS; Dopamine; PET

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active tDCS (Active Comparator): Intensity : 2mA Duration : 20 minutes ramp up/ramp down 30sec anodal tDCS applied over the left DLPFC cathodal tDCS applied over the right DLPFC
  Interventions: Device: Procedure: active tDCS
- sham tDCS (Placebo Comparator): Placebo built-in mode (30 sec ramp periods at the beginning and the end of the sham stimulation to mimic the somatosensory artifact of real tDCS) Same electrode montage than in the active group.
  Interventions: Device: Procedure: sham tDCS

INTERVENTIONS:
Device: Procedure: active tDCS — Intensity 2 mA during 20 minutes
  Arms: active tDCS
Device: Procedure: sham tDCS — sham condition as delivered by the stimulator
  Other Names: tDCS placebo
  Arms: sham tDCS

SUMMARY:
Transcranial direct current stimulation (tDCS) is a technique that is emerging as a prospective therapy for neurologic, psychiatric and addictive disorders. Specifically, anodal tDCS applied over the dorsolateral prefrontal cortex (DLPFC) is associated with improvement of cognitive functions and mood. Despite an increased use in clinical settings, tDCS suffers from limitations, especially regarding the strength and the duration of therapeutic effects. Strategies to optimize the conditions for tDCS application suffer from the lack of knowledge about its neurophysiological impact. Moreover, tDCS is increasingly used in private settings through commercial apparatus and tutorials to make a "do-it-yourself" device delivering tDCS now available on the Internet. This private use worries neuroscientists and health authorities. Even if the general impression is that, in controlled conditions, tDCS is safe with only mild and transient adverse effects, whether and how tDCS could be used for enhancing cognition in healthy subjects are needed to investigate in more detail. The investigators believe that a better understanding of some neurobiological effects of tDCS is crucial to further tailor tDCS for experimental and therapeutic applications and to define recommendations for a private use.

As the cortex is densely connected with basal ganglia areas, including dopaminergic areas, tDCS is probably not only capable to target cortical but also subcortical structures remote from the stimulation sites. Some studies suggest that cortical stimulation by other approaches, such as transcranial magnetic stimulation (rTMS) leads to an increased dopaminergic transmission. The involvement of dopaminergic systems in tDCS effects has been investigated only indirectly in pharmacological studies. Thus, the direct effect of the DLPFC stimulation by tDCS on dopaminergic transmission is still unknown.

The aim of this project is to reveal the online impact of a single-session of tDCS applied bilaterally over the DLPFC in healthy subjects on the dopaminergic transmission measured by PET, combined with the [11C]raclopride bolus-plus-continuous-infusion method.

ELIGIBILITY:
Inclusion Criteria:

* Non smoker
* No pyschotrope consumption
* No medical treatment
* No psychiatric or somatic (neurological, endocrine, cardiac, renal)
* Affiliated to the french social security

Exclusion Criteria:

* No consent
* For females : Pregnant or without birth control
* Contraindications to stimulation by tDCS or to an MRI exam
* Being in an exclusion period or over the annual compensation ceiling
* Participation in another study using ionizing radiation in less than a year

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in dopamine transmission after 1 session of 20min tDCS | during 100min of PET scan : Baseline (20-40min), during stimulation (40-60min) and after stimulation (60-80min & 80-100min)
  Measure of the Binding Ratio defined as the ratio of : region of interest / cerebellum activities)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Haesebaert, PH, Principal Investigator — CH Le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, France